CLINICAL TRIAL: NCT00771784
Title: Effects of Short- and of Long-term Tracheal Intubation on Ventilation With a Laryngeal Mask During Percutaneous Dilatation Tracheostomy.
Brief Title: Effects of Tracheal Intubation on Ventilation With a Laryngeal Mask During Percutaneous Dilatation Tracheostomy
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Michele Carron/MD, Department of Pharmacology and Anesthesiology, University of Padova
Other Study IDs: 68144
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Neurological Diseases, Heart or Respiratory Failure,; Sepsis, Trauma.
Keywords: Endotracheal intubation; tracheostomy; laryngeal mask
MeSH Terms: conditions — Respiratory Insufficiency; Sepsis; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Short term endotracheal intubation.
- 2: Long term endotracheal intubation.

SUMMARY:
The length of tracheal intubation may affect the subsequent ventilation with a laryngeal mask during percutaneous tracheostomy.

DETAILED DESCRIPTION:
Percutaneous tracheostomy is routinely performed while patients are being ventilated with a laryngeal mask. The efficacy of ventilation during tracheostomy may be affected by length of previous endotracheal intubation.

This is an observational and monocentric study aimed to evaluate the impact of length of endotracheal intubation on efficacy of lung ventilation with a laryngeal mask. Two groups of patients who have to undergo elective percutaneous tracheostomy after either a short or long endotracheal intubation will be enrolled.

Data on the correlational effects of the endotracheal tube on the integrity of laryngeal structures and on ventilation will be collected.

Statistical analyses will use standard tests to compare the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* mechanical ventilation
* need of percutaneous tracheostomy

Exclusion Criteria:

* previous pathologies of upper airways or of oesophagus
* risk of bleeding
* need of FiO2 >70% and/or of PEEP >10 cm H2O
* difficult insertion of laryngeal mask
* impossibility of endoscopic visualization of the laryngeal structures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Ventilatory parameters during percutaneous tracheostomy | Thirty minutes.

SECONDARY OUTCOMES:
Scoring of laryngeal lesions, blood gas exchange, morbidity, mortality. | Thirty minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ori, Professor, Study Chair — Department of Pharmacology and Anesthesiology, University of Padova
Locations (1):
- Intensive Care Unit, S. Anthony Hospital, Padua, PD, Italy

REFERENCES:
- See also: Link of the Anesthesia and Critical Care Section — http://www.istar.unipd.it/